CLINICAL TRIAL: NCT03044470
Title: Role of Cryotherapy in Reduction of Post Operative Endodontic Pain Following Single Visit Root Canal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mamata Dental College (Other)
Responsible Party: Principal Investigator, KIRIT GOLLA, POST GRADUATE, Mamata Dental College
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mamata DC
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Effects of; Cold
MeSH Terms: conditions — Common Cold | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold saline (Experimental): Saline stored at 4 degrees centigrade
  Interventions: Other: cryotherapy
- Normal Saline (Experimental): Saline stored at room temperature
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: cryotherapy — Role of cryotherapy in reduction of post operative pain
  Other Names: Cold saline

SUMMARY:
AIM : To determine the efficacy of cold saline irrigation in reduction of post operative pain following root canal therapy.

METHODOLOGY : Forty patients requiring root canal treatment on permanent single rooted teeth were included. The patients were assigned randomly into two groups of 20 patients each. The teeth in Group1 (n = 20) were irrigated using normal saline solution, whilst those in Group 2 (n = 20) were irrigated with cold saline solution stored at 4 degrees centigrade. A Heft Parker visual analog scale was used to measure pre-operative pain and post-obturation pain at 12, 24,48 and 72 hours after obturation. Chi square tests and Mann Whitney U tests were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Healthy patients without any medical conditions

Exclusion Criteria:

* root canal retreatment
* pregnancy
* teeth with open apices
* a history of intolerance to nonsteroidal anti-inflammatory drugs
* immunosuppressed patients
* those under 18 years old
* patients requiring antibiotic prophylaxis
* patients with pacemakers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-09-05 (Actual)

PRIMARY OUTCOMES:
Post endodontic pain measure at different time intervals using heft parker visual analog scale | 12,24,48,72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mamata Dental College, Khammam, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided